CLINICAL TRIAL: NCT01869634
Title: Mechanisms of Immune Reconstitution & Reduced Immune Activation Following Darunavir-based ART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 394080; IIS RFA _Asmuth:TMC114HIV2029 (Other: Other)
Record Dates: First submitted 2013-06-01; First posted 2013-06-05 (Estimated); Results first posted 2020-03-04 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-02

CONDITIONS: Human Immunodeficiency Virus Infection
Keywords: HIV; cardiovascular risk; systemic immune activation
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIV positive naive to ART (Active Comparator): HIV subjects will receive open-label darunavir 800 mg in combination with ritonavir 100 mg tablets and fixed-dose combination viread + emtricitabine (Truvada®) to be taken once daily without regard to food. Subjects will undergo upper endoscopy, CT cardiac angiogram, intimal-medial thickening, and peripheral blood collection before and after 12 months of ART.
  Interventions: Drug: darunavir with ritonavir and fixed-dose viread+emtricitabine daily
- normal control volunteers (No Intervention): HIV negative age-matched controls will undergo the same interventions and procedures without receiving ART at study entry and after 12 months.

INTERVENTIONS:
Drug: darunavir with ritonavir and fixed-dose viread+emtricitabine daily
  Other Names: darunavir (Prezista®) 800 mg with ritonavir 100 mg and Truvada® to be taken once daily
  Arms: HIV positive naive to ART

SUMMARY:
Potent HIV suppression with Darunavir-based antiretroviral therapy (ART) will lead to repopulation of gastrointestinal-associated lymphoid tissue (GALT) cluster of differentiation (CD)4+ T-cell populations, normalization of systemic immune activation, and improved HIV-associated cardiovascular disease (CVD) risk.

DETAILED DESCRIPTION:
Rationale Infection with HIV causes significant morbidity and mortality, even among individuals who are virologically suppressed with combination anti-retroviral therapy (ART). ART is effective in prolonging life and enabling individuals who are HIV positive to live near-normal life spans. However, these individuals are increasingly developing a number of chronic diseases of aging, such as atherosclerotic cardiovascular disease (ASCVD). The proposed studies will examine the role of highly active antiretroviral therapy in restoring the mucosal immunity and the systemic effect on immune activation, bacterial translocation, and change in HIV-associated cardiovascular disease risk.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign consent form
* Naïve to ART (remote ART use >5 years will be considered on a case by case basis)
* No known GI or cardiovascular disease
* Between the ages of 18 and 60
* No active opportunistic infections or therapy for acute OI within 30 days of entry. Subjects can be on secondary prophylaxis with a history of AIDS defining illness.
* All women of childbearing potential (WCBP) must have a negative urine pregnancy test before any of the invasive or radiation exposure study procedures.
* Normal population should be free of chronic metabolic conditions such as diabetes, hypercholesterolemia, or coronary artery disease
* There are no CD4+ T-cell count or HIV plasma viral load restrictions.

Exclusion Criteria:

* Abnormal coagulation parameters (PT>1.2 upper limit of normal (ULN))
* Thrombocytopenia (platelet count <50.000 within 6 weeks)
* Contra-indications to upper endoscopy or conscious sedation
* Anemia (>grade 1 [appendix 1])
* Aspirin, ibuprofen, warfarin or other agents that interfere with the coagulation cascade are prohibited within 1 week of endoscopy.
* Renal insufficiency (serum Creatinine >1.2 ULN)
* History of chronic proteinuria that could impact viread use.
* Allergy to contrast used for CT angiography
* Requirement to take medications that are contraindicated with study ART regimen.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- HIV Positive Naive to ART: HIV subjects will receive open-label darunavir 800 mg in combination with ritonavir 100 mg tablets and fixed-dose combination viread + emtricitabine (Truvada®) to be taken once daily without regard to food. Subjects will undergo upper endoscopy, CT cardiac angiogram, intimal-medial thickening, and peripheral blood collection before and after 12 months of ART.
  darunavir with ritonavir and fixed-dose viread+emtricitabine daily
Period: Overall Study
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers
Started | 20 | 17
Completed | 18 | 17
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 17 | 35
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 40 [31 to 51] | 37 [33 to 47] | 37 [32 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 18 | 17 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 2 | 6
  White | 7 | 8 | 15
  More than one race | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 17 | 35
CD4+ T-cells [Median (Inter-Quartile Range); unit: cells/mm^3] | 215 [150 to 260] | 460 [370 to 530] | 310 [210 to 460]
HIV viral load [Median (Inter-Quartile Range); unit: copies/ml] | 41032 [20689 to 78805] | 0 [0 to 0] | 41032 [20689 to 78805]
weight [Median (Inter-Quartile Range); unit: lbs] | 187 [153 to 200] | 194 [176 to 210] | 191 [170 to 210]

OUTCOME MEASURES:

1. Primary Outcome: Number of CD4+ T-cells in the Lamina Propria/mm2 Before and After 12 Months of Therapy Compared to Age-matched Control Volunteers Without HIV
Description: CD4+ T-cells in the lamina propria/mm2 before and after 12 months of therapy compared to age-matched control volunteers without HIV.
Time Frame: Baseline, 12 months
Population: HIV negative participants underwent the procedures only once at Screening (entry). In the HIV group the comparison between before and after ART was done using a Wilcoxon signed-rank test.
Measure: Median (Inter-Quartile Range); unit: cells / mm^2
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers
Number analyzed (Participants) | 18 | 17
cells / mm^2
  Entry | 80 [34 to 190] | 478 [389 to 627]
  12-months after ART: number analyzed (Participants) | 18 | 0
  12-months after ART | 213 [120 to 292] |
Statistical Analysis 1: Comparison: HIV Positive Naive to ART; Comparison between HIV positive naïve to ART before and after ART has been done; Test type: Other — Wilcoxon signed-rank test. Paired samples; p = 0.0025, Sign test

2. Secondary Outcome: Change in Percentage of Total Artery Diameter
Description: computerized axial tomography angiography of the coronary arteries (CT-angio) before and after 12-months of Darunavir therapy
Time Frame: Baseline, 12 months
Population: We compare wall thickness between HIV+ infected individuals and in the HIV group before and after 12-months of ART.
Measure: Median (Inter-Quartile Range); unit: % of total artery diameter
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers
Number analyzed (Participants) | 15 | 14
% of total artery diameter | 57 [54 to 61] | 53 [50 to 56]
Statistical Analysis 1: Comparison: HIV Positive Naive to ART vs Normal Control Volunteers; Test type: Other — Two-sample Wilcoxon rank-sum (Mann-Whitney) test; p = 0.032, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: HIV Positive Naive to ART; Comparison of coronary artery wall thickness before and after ART in the HIV infected participants; Test type: Other — Wilcoxon signed-rank test; p = 0.826, Sign test

3. Other Pre Specified Outcome: Change in Systemic Immune Activation
Description: Change in systemic immune activation, as measured by change in plasma cytokine levels (IL-6).
Time Frame: Baseline, 12 months
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers
Number analyzed (Participants) | 18 | 17
pg/ml | 1.74 [1.42 to 2.15] | 0.66 [0.50 to 0.81]
Statistical Analysis 1: Comparison: HIV Positive Naive to ART vs Normal Control Volunteers; comparison between groups (HIV+ vs HIV-); Test type: Other — Two-sample Wilcoxon rank-sum (Mann-Whitney) test; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: HIV Positive Naive to ART; Changes in systemic immune activation through IL6; Test type: Other; p = 0.807, Sign test

ADVERSE EVENTS:
Arm/Group | HIV Positive Naive to ART | Normal Control Volunteers
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes